CLINICAL TRIAL: NCT01127893
Title: A PHASE 3, MULTICENTER, RANDOMIZED, LONG TERM STUDY OF THE SAFETY OF THE SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN PATIENTS WITH OSTEOARTHRITIS OF THE KNEE
Brief Title: Safety Extension Study Of Tanezumab When Administered By Subcutaneous Injection To Patients With Osteoarthritis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091032; SAFETY EXTENSION OF 1027 (Other: Alias Study Number)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Osteoarthritis
Keywords: Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis; Musculoskeletal Diseases; Joint Diseases; Arthritis; Rheumatic Diseases | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tanezumab 10 mg (Experimental)
  Interventions: Biological: Tanezumab
- Tanezumab 5 mg (Experimental)
  Interventions: Biological: Tanezumab
- Tanezumab 2.5 mg (Experimental)
  Interventions: Biological: Tanezumab

INTERVENTIONS:
Biological: Tanezumab — Tanezumab 10 mg administered by subcutaneous injection every 8 weeks for up to 7 injections
  Arms: Tanezumab 10 mg
Biological: Tanezumab — Tanezumab 5 mg administered by subcutaneous injection every 8 weeks for up to 7 injections
  Arms: Tanezumab 5 mg
Biological: Tanezumab — Tanezumab 2.5 mg administered by subcutaneous injection every 8 weeks for up to 7 injections
  Arms: Tanezumab 2.5 mg

SUMMARY:
An evaluation of the long term safety of tanezumab when administered by subcutaneous injection every 8 weeks for up to 64 weeks

DETAILED DESCRIPTION:
This study was terminated on 29 September 2010 following a US FDA clinical hold for tanezumab osteoarthritis clinical studies which halted dosing and enrollment of patients on 23 June 2010 for potential safety issues.

ELIGIBILITY:
Inclusion Criteria:

* Must have participated in specific Phase 3 parent study

Exclusion Criteria:

* Failed screening for parent study, pregnant women, lactating mothers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06-15 (Actual); Primary Completion 2010-09-29 (Actual); Study Completion 2010-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Triwest Research Associates, La Mesa, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4091032&StudyName=Safety%20Extension%20Study%20Of%20Tanezumab%20When%20Administered%20By%20Subcutaneous%20Injection%20To%20Patients%20With%20Osteoarthritis%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had received tanezumab 2.5 milligram(mg) subcutaneously(SC) every 8 weeks, 5 mg SC every 8 weeks or 10 mg SC or intravenously every 8 weeks in parent Study A4091027 (NCT01089725) were to be assigned to same dose group and who received placebo in same parent study, were to be randomized to either tanezumab 2.5, 5 or 10 mg SC every 8 weeks in this study.
Pre-assignment Details: Due to the United States Food and Drug Administration (US FDA) imposed clinical hold, the study was terminated prematurely. Only 1 participant was enrolled and treated with tanezumab 2.5 mg treatment group and other planned treatments, tanezumab 5 or 10 mg, were not administered.
Groups:
- Tanezumab 2.5 mg: Participants who had previously received tanezumab (RN624 or PF-04383119) 2.5 mg subcutaneous injection every 8 weeks in parent Study A4091027 (NCT01089725), received single dose of tanezumab 2.5 mg subcutaneous injection on Day 1.
Period: Overall Study
Arm/Group | Tanezumab 2.5 mg
Started | 1
Completed | 0
Not Completed | 1
Not completed — Study Termination by the Sponsor | 1

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) analysis population included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug, up to early termination (Day 107) that were absent before treatment in this study or that worsened relative to pretreatment state.
Time Frame: Baseline up to Early Termination (Day 107)
Population: ITT analysis population included all randomized participants who received at least 1 dose of study medication. Due to the US FDA imposed clinical hold, the study was terminated prematurely. Consequently, all planned analyses were not performed; data reported here is for baseline up to early termination (Day 107).
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants
  AEs | 0
  SAEs | 0

2. Primary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Laboratory examination included blood chemistry, hematology and urinalysis. Reported results were to include abnormal laboratory findings without regard to baseline abnormality.
Time Frame: Baseline up to Early Termination (Day 107)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants | 0

3. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Following parameters were analyzed for ECG abnormality: PR interval, QRS interval, QT interval, QT interval corrected using the Bazett's formula (QTcB), QT interval corrected using Fredericia's formula (QTcF), RR interval and heart rate (HR).
Time Frame: Baseline up to Early Termination (Day 107)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants | 0

4. Primary Outcome: Number of Participants With Neurologic Examination Abnormalities
Description: Neurologic examination assessed the strength of groups of muscles of the head and neck, upper limbs and lower limbs, deep tendon reflexes and sensation (tactile, vibration, joint position sense and pin prick) of index fingers and great toes.
Time Frame: Baseline up to Early Termination (Day 107)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants | 0

5. Primary Outcome: Number of Participants With Anti-Drug (Tanezumab) Antibody (ADA)
Description: Human serum ADA samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline up to Early Termination (Day 107)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants | 0

6. Primary Outcome: Number of Participants With Injection Site Reactions
Description: Injection site reactions included: erythema (redness), induration (swelling), ecchymosis (bruising), pruritus (itching) and pain that occurred after the injection has been administered.
Time Frame: Baseline up to Early Termination (Day 107)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants | 0

7. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint in the past 48 hours. It is calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicated higher pain. Total score range for WOMAC pain subscale score is 0 to 10, where higher scores indicated higher pain.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: ITT analysis population included all randomized participants who received at least 1 dose of study medication. Due to the US FDA imposed clinical hold, only 1 participant was enrolled and the study was terminated prematurely. Consequently, planned analyses for Week 8, 16, 24, 32, 40, 48, 56, and 64 were not performed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 5.8
  Change at Week 4 | 0.0

8. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale Score at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: The WOMAC physical function subscale is a 17-item questionnaire used to assess the degree of difficulty experienced due to osteoarthritis in the index joint in the past 48 hours. It is calculated as the mean of the scores from the 17 individual questions scored on a NRS of 0 to 10, where higher scores indicated worse function. Total score range for WOMAC physical function subscale score is 0 to 10, where higher scores indicate worse function. Physical function refers to participant's ability to move around and perform usual activities of daily living.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 6.2
  Change at Week 4 | -0.1

9. Secondary Outcome: Change From Baseline in Patient Global Assessment (PGA) of Osteoarthritis at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: PGA: Participants answered the following question: "Considering all the ways your osteoarthritis (OA) in your knee affects you, how are you doing today?" Participants rated their condition by using a 5-point Likert scale: 1) Very Good (asymptomatic and no limitation of normal activities); 2) Good (mild symptoms and no limitation of normal activities); 3) Fair (moderate symptoms and limitation of some normal activities); 4) Poor (severe symptoms and inability to carry out most normal activities); and 5) Very Poor (very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 3.0
  Change at Week 4 | 0.0

10. Secondary Outcome: Percentage of Participants With Outcome Measures in Rheumatoid Arthritis Clinical Trials - Osteoarthritis Research Society International (OMERACT-OARSI) Response
Description: OMERACT-OARSI response: >=50 percent (%) improvement from baseline and absolute change from baseline of >=2 units at Week of interest in WOMAC pain or physical function subscale, or at least 2 of the following 3 being true: >=20% improvement from baseline and absolute change from baseline of >=1 unit at Week of interest in 1) WOMAC pain subscale, 2) WOMAC physical function subscale, 3) PGA of osteoarthritis (score: 1-5, higher score=more affected). WOMAC pain, physical function subscales assess amount of pain/difficulty experienced (score: 0-10, higher score=higher pain/difficulty).
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: Due to the US FDA imposed clinical hold, only 1 participant was enrolled and the study was terminated prematurely. Consequently, planned efficacy analysis was not performed.
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants With At Least 30 Percent (%), 50%, 70% and 90% Reduction in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: The WOMAC pain subscale is a 5-item questionnaire used to assess the amount of pain experienced due to osteoarthritis in the index joint in the past 48 hours. It was calculated as the mean of the scores from the 5 individual questions scored on a numerical rating scale (NRS) of 0 to 10, where higher scores indicated higher pain. Total score range for WOMAC pain subscale score was 0 to 10, where higher scores indicated higher pain.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 10
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Cumulative Reduction From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score
Description: as for outcome 11
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 10
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Participants With Improvement of At Least (>=) 2 Point in Patient Global Assessment (PGA) of Osteoarthritis
Description: PGA: Participants answered the following question: "Considering all the ways your OA in your joint affects you, how are you doing today?" Participants rated their condition by using a 5-point Likert scale: 1) Very Good (asymptomatic and no limitation of normal activities); 2) Good (mild symptoms and no limitation of normal activities); 3) Fair (moderate symptoms and limitation of some normal activities); 4) Poor (severe symptoms and inability to carry out most normal activities); and 5) Very Poor (very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 10
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Stiffness Subscale Score at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: The WOMAC stiffness subscale is a 2-item questionnaire used to assess the amount of stiffness experienced in the index joint in the past 48 hours. It was calculated as the mean of the scores from the 2 individual questions scored on NRS of 0 to 10; where higher scores indicated more stiffness. Total score range for WOMAC stiffness subscale score is 0 to 10, where higher scores indicated more stiffness. Stiffness is defined as a sensation of decreased ease in movement of the index joint.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 6.5
  Change at Week 4 | 0.0

15. Secondary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Average Score at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: WOMAC: self-administered, disease-specific 24-item questionnaire which assesses clinically important, participant-relevant symptoms for pain (5 items), stiffness (2 items) and physical function (17 items) in participants with osteoarthritis. WOMAC average score was the mean of WOMAC pain, physical function and stiffness subscale scores and ranges from 0 to 10, where higher score indicated worse response.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 6.2
  Change at Week 4 | -0.1

16. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item (Pain When Walking on a Flat Surface) at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: Participants answered: "How much pain have you had when walking on a flat surface?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 5.0
  Change at Week 4 | 0.0

17. Secondary Outcome: Change From Baseline in WOMAC Pain Subscale Item (Pain When Going Up or Down Stairs) at Week 4, 8, 16, 24, 32, 40, 48, 56, and 64
Description: Participants answered: "How much pain have you had when going up or down stairs?" Participants responded by using a NRS of 0 to 10, where 0 = no pain and 10 = extreme pain.
Time Frame: Baseline, Week 4, 8, 16, 24, 32, 40, 48, 56, 64
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
units on a scale
  Baseline | 7.0
  Change at Week 4 | 0.0

18. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Time Frame: Baseline up to Week 64
Population: Data not analyzed since no participant discontinued the study due to lack of efficacy.
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants Who Received Concomitant Analgesic Medication for Osteoarthritis Treatment
Description: Permissible concomitant analgesic medications included Food and Drug Administration (FDA) approved opioids, topical analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), capsaicin products, oral/injectable corticosteroids and viscosupplementation (for example, hyaluronan) and were to be prescribed as per investigator's discretion.
Time Frame: Baseline up to Day 107 (Early Termination)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
Participants | 0

20. Secondary Outcome: Days Per Week of Concomitant Analgesic Medication Usage for Osteoarthritis Treatment
Description: as for outcome 19
Time Frame: Baseline up to Week 64
Population: Data not analyzed since no participant received concomitant analgesic medication.
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 0

21. Secondary Outcome: Tanezumab Plasma Concentration
Time Frame: Pre-dose on Week 8, 24, 40; Week 56, 64
Population: ITT analysis population included all randomized participants who received at least 1 dose of study medication. Due to the US FDA imposed clinical hold, the study was terminated prematurely (Day 107). Consequently, planned analyses for Week 24, 40, 56 and 64 were not performed.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
nanogram per milliliter (ng/mL)
  Week 8 | 63.7
  Early Termination (Day 107) | NA — Data not reported since the observed concentration was below lower limit of quantification (12 ng/mL).

22. Secondary Outcome: Nerve Growth Factor (NGF) Serum Concentration
Description: Serum samples were analyzed for determining total NGF concentration. Total NGF was analyzed using a validated, sensitive, and specific immune-affinity enrichment liquid chromatography tandem mass spectrometric (IA/LC/MS/MS) method.
Time Frame: Pre-dose on Week 8, 24, 40; Week 56, 64
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Tanezumab 2.5 mg
Number analyzed (Participants) | 1
picogram per milliliter (pg/mL)
  Week 8 | 1138
  Early Termination (Day 107) | 208.9

ADVERSE EVENTS:
Arm/Group | Tanezumab 2.5 mg
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Due to the US FDA imposed clinical hold, enrollment and further dosing with study medication was stopped prematurely, only 1 participant was enrolled and the study was terminated early. Designation of outcomes as primary, secondary based on study team input as study did not specify them as primary or secondary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.